CLINICAL TRIAL: NCT00302575
Title: Step'n Out: A Multisite Trial of Collaborative Behavioral Management for Drug-Involved Parolees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Collaborators: Substance Abuse and Mental Health Services Administration (SAMHSA) (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1U01DA016191 (NIH)
Record Dates: First submitted 2006-03-13; First posted 2006-03-14 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2006-08

CONDITIONS: Substance-Related Disorders
Keywords: Substance-Related Disorders; Prisoners
MeSH Terms: conditions — Substance-Related Disorders

INTERVENTIONS:
Behavioral: Collaborative Behavioral Management
Procedure: Integrated parole and outpatient addiction treatment

SUMMARY:
The main purpose of this study is to examine whether improved integration between the community supervision system and outpatient addiction treatment system can improve treatment adherence, drug use and public safety outcomes among drug-involved inmates re-entering the community.

DETAILED DESCRIPTION:
The target population consists of male and female parolees with a history of substance abuse treatment who are at moderate-to-high-risk of recidivism. They will recruited from in the criminal justice system and/or transitional residential drug treatment within one or two months of release or at the time they first report for parole supervision.

Participants from six states (KY, OR, RI, CT, VA, DE) will be randomized into the Step'n Out condition (integration of community supervision and addiction treatment with behavioral management) or a comparison condition including traditional community supervision and addiction treatment. Research interviews at baseline, and 3 and 9 months after release from confinement will assess study participants' outcomes.

The Step'n Out intervention will produce significantly better outcomes than the standard referral condition with respect to: recidivism rates (revocation, rearrest on a new charge, reconviction, reincarceration), as assessed 3 and 9 months after the end of the intervention; treatment participation (i.e., proportion of planned sessions attended, proportion of planned days retained in treatment, type of discharge [successful completion, transfer to another program, elopement, administrative discharge, return to custody], as assessed after the end of the intervention; self-reported drug use, criminal activity, and psychosocial functioning, as assessed 3 and 12 months after the end of the intervention; cost-effectiveness; collaboration between the supervision officer and treatment counselor ; and therapeutic alliance with the clients.

ELIGIBILITY:
Inclusion Criteria:

1. be at least 18 years old and speak English;
2. have probable drug dependence immediately prior to incarceration as determined by a score of 3 or higher on the TCU Drug Screen II;
3. be at moderate-to-high-risk of drug relapse and/or recidivism as determined by a Lifestyle Criminality Screening Form (LCSF) score of 7 or greater, or a history of 2 or greater prior treatments for drug-related problems or drug-related convictions;
4. must have substance use treatment as a mandated or recommended condition of parole.

Exclusion Criteria:

1. psychotic features;
2. parole or probation conditions that prohibit them from participating in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2005-02; Study Completion 2007-08 (Estimated)

PRIMARY OUTCOMES:
Rearrest

SECONDARY OUTCOMES:
Drug use

CONTACTS AND LOCATIONS:
Overall Officials: Peter D Friedmann, MD, MPH, Principal Investigator — Rhode Island Hospital
Locations (5):
- United States (5):
  - University of California, Los Angeles, Los Angeles, California
  - Connecticut Deptartment of Mental Health & Addiction Services, Hartford, Connecticut
  - University of Delaware, Newark, Delaware
  - University of Kentucky, Lexington, Kentucky
  - Virginia Commonwealth University, Richmond, Virginia

REFERENCES:
- [Derived] Friedmann PD, Green TC, Taxman FS, Harrington M, Rhodes AG, Katz E, O'Connell D, Martin SS, Frisman LK, Litt M, Burdon W, Clarke JG, Fletcher BW; Step'n Out Research Group of CJ-DATS. Collaborative behavioral management among parolees: drug use, crime and re-arrest in the Step'n Out randomized trial. Addiction. 2012 Jun;107(6):1099-108. doi: 10.1111/j.1360-0443.2011.03769.x. Epub 2012 Feb 28. PMID 22175445